CLINICAL TRIAL: NCT06296485
Title: Pragmatic Clinical Trial of Continuous Glucose Monitoring-based Interventions for Safe Insulin Use in High-Risk Older Adults With Type 2 Diabetes
Brief Title: Safer Aging With Diabetes Monitoring
Acronym: SAGE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB-1996616; R01DK134446 (NIH)
Record Dates: First submitted 2024-02-29; First posted 2024-03-06 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2024-10

CONDITIONS: Diabetes Mellitus, Type 2; Hypoglycemia
Keywords: Hypoglycemia; Diabetes Education; Continuous Glucose Monitor
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypoglycemia

STUDY DESIGN:
Intervention Model Description: 2-arm pragmatic randomized clinical trial
Who Masked: Outcomes Assessor
Masking Description: Participant randomization status will be masked during data collection (baseline and follow-up surveys) by research assistants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Education Sessions (Experimental): Participants will participate in 3 educational sessions designed to teach about applying and using continuous glucose monitors [CGMs] (Session 1) and how to prevent hypoglycemia episodes based on CGM readings and hypoglycemia journal entries (Sessions 2 & 3).
  Interventions: Behavioral: SAGE Group Sessions
- Usual Care (Active Comparator): Participants allocated to the control arm will continue with usual care.
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: SAGE Group Sessions — Participants enroll in 3 educational group sessions and receive CGMs
  Arms: Group Education Sessions
Other: Usual Care — Participants continue to receive usual care (Control Arm)
  Arms: Usual Care

SUMMARY:
Older adults with type 2 diabetes are at higher risk for severe hypoglycemia and its related complications (including hospitalization and death) when taking insulin. This study proposes to evaluate, in a randomized clinical trial, a strategy of safe insulin prescribing based on an educational program that leverages continuous glucose monitoring to support older adults at high risk for hypoglycemia. If the aims of this project are achieved, this novel care strategy could be widely applied to reduce severe hypoglycemia episodes in older, high-risk adults with type 2 diabetes.

DETAILED DESCRIPTION:
The overarching goal of this pragmatic randomized clinical trial is to support safer diabetes care in older adults (age ≥ 75) with type 2 diabetes (T2D) who require insulin therapy. Many of these older adults are at high risk for severe hypoglycemia due to symptom unawareness and/or nocturnal hypoglycemia. Effective and safe management in this population requires close glucose monitoring coupled with proactive medication and diet adjustment to avoid severe iatrogenic consequences. This study proposes to achieve this goal through a patient-oriented intervention program that incorporates the use of alarm-enabled continuous glucose monitoring (CGM). There are currently no major randomized trials directly assessing the use of CGM to reduce severe hypoglycemia among the oldest adults with T2D. The study team will conduct a 2-arm trial: 1) Group-based, three-session education intervention (CGM provided to participants) vs. 2) usual care (no CGM provided to participants). The primary outcome is an aggregate measure of clinically significant hypoglycemia. The study will also examine differences in patient-reported diabetes distress, fear of hypoglycemia, and self-efficacy using validated survey measures.

ELIGIBILITY:
Inclusion Criteria:

* Age 75 years and older
* Diagnosis of Type 2 Diabetes
* Current treatment with insulin
* Increased hypoglycemia risk (prior year hypoglycemia by self-report or utilization)
* Able to communicate in English
* Able to access email and the Internet

Exclusion Criteria:

* On renal dialysis
* Dementia
* Pacemaker or Automatic Implantable Cardioverter Defibrillator
* Using insulin pump
* Severe Mental Illness
* Severe Visual Impairment
* In Hospice
* Current or recent CGM use

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2027-03-30 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Hypoglycemia aggregate outcome | 6 and 12 months after study start date
  This outcome will compare the proportion of patients in the three study arms with self-reported hypoglycemia (symptomatic and/or requiring help from others) and/or hypoglycemia-related utilization (emergency department, hospital or outpatient new events) 6- and 12-months after enrollment

SECONDARY OUTCOMES:
Self-reported hypoglycemia | 6 and 12 months after study start date
  This outcome will compare the proportion of patients in the three study arms with self-reported hypoglycemia (symptomatic and/or requiring help from others)
Hypoglycemia-related utilization | 6 and 12 months after study start date
  This outcome will compare the proportion of patients in the three study arms with hypoglycemia-related utilization (emergency department, hospital or outpatient new events)
Diabetes Distress | 6 and 12 months after study start date
  This outcome will compare responses to the 2-item, validated Diabetes Distress survey
Hypoglycemia Confidence | 6 and 12 months after study start date
  This outcome will compare responses to the 9-item, validated Hypoglycemia Confidence survey
Hypoglycemia Distress | 6 and 12 months after study start date
  This outcome will compare responses to the 3-item, validated Hypoglycemia Distress survey

OTHER OUTCOMES:
Technology Proficiency | 6 and 12 months after study start date
  This outcome will compare responses to a 3-item subset of the validated Technology Proficiency survey
Confidence in Adjusting Insulin | 6 and 12 months after study start date
  This outcome will assess confidence in adjusting insulin across the 3 study arms using a 3-item survey
Insulin Adjustment | 6 and 12 months after study start date
  This outcome will assess patient self-report of changes to insulin regimen in preceding 6 months
Caregiver Action | 6 and 12 months after study start date
  This outcome will assess patient self-report of caregiver taking action to address low blood sugar in preceding 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Richard W Grant, MD MPH, Principal Investigator — Kaiser Permanente Northern California - Division of Research
Locations (4):
- United States (4):
  - Kaiser Permanente Fremont, Fremont, California
  - Kaiser Permanente San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Kaiser Permanente - Union City, Union City, California

IPD SHARING:
Plan to Share IPD: No